CLINICAL TRIAL: NCT04211961
Title: A Randomised Double-Blinded Placebo-Controlled Trial to Assess the Efficacy and Safety of Scopolamine Compared to Placebo in Individuals With Bipolar Disorder Who Are Experiencing a Depressive Episode
Brief Title: Scopolamine in Bipolar Depression
Acronym: SCOPE-BD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Brian Hallahan (Other)
Collaborators: Stanley Medical Research Institute (Other); National University of Ireland, Galway, Ireland (Other); HRB Clinical Research Facility Galway (Other); University College Hospital Galway (Other)
Responsible Party: Sponsor-Investigator, Dr. Brian Hallahan, Senior Lecturer and Consultant Psychiatrist, Department of Psychiatry, National University of Ireland, Galway, Ireland
Organization: National University of Ireland, Galway, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUIG-2017-002; 2017-003112-39 (EudraCT Number)
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Disorder Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Sodium Chloride; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants randomised to the placebo group will receive one 15-minute IV infusion of 100ml Saline at 4 visits.
  Interventions: Other: Placebo / Saline
- Scopolamine (Active Comparator): Participants randomised to the Scopolamine/treatment group will receive one 15-minute IV infusion of Scopolamine at 4 visits.
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Other: Placebo / Saline — The placebo group will receive a 100ml infusion of saline at 4 visits during the study
  Arms: Placebo
Drug: Scopolamine — The treatment group will receive a 100ml infusion of Scopolamine ( dose 4μg/kg) at 4 visits during the study
  Arms: Scopolamine

SUMMARY:
This is a single-site, randomised, double-blind, placebo-controlled, parallel, phase IIb clinical trial. The primary objective of the SCOPE-BD study is to investigate the efficacy and safety of IV Scopolamine, compared to placebo, in reducing severity of depression in individuals with bipolar disorder who are experiencing a depressive episode of at least moderate severity

DETAILED DESCRIPTION:
Bipolar disorder is a chronic disabling psychiatric disorder characterized by recurrent episodes of mania or hypomania and depression. Bipolar disorder can be separated into bipolar 1 and bipolar 2 disorders with bipolar 1 disorder characterizing individuals who have episodes of mania and depression, and bipolar 2 disorder characterizing individuals who have episodes of depression with periods of hypomania, but not mania. Bipolar disorder has an estimated prevalence of approximately 1% and a roughly equal gender ratio. Current pharmacological treatments for bipolar disorder and in particular for the management of depressive episodes in bipolar disorder remain sub-optimal, with pharmacological strategies employed to date often only partially effective. In addition to the time duration for treatment response, multiple treatment trials are also often required, thus increasing patient discomfort and distress.Consequently, pharmacological mechanisms that potentially alleviate depressive symptomatology in bipolar disorder and ameliorate patient functioning could present an additional pharmacological strategy for the management of bipolar disorder. A number of recent studies have suggested that Scopolamine, a pan muscarinic (M) receptor antagonist can elicit a rapid anti-depressant response in both major depressive disorder (MDD) and bipolar disorder and thus may present a novel therapeutic strategy, particularly for the management of bipolar disorder, in individuals experiencing depressive episodes. No significant adverse effects were noted with treatment with Scopolamine (intravenously) in these studies.

This antidepressant effect has been rapid in effect in studies where administration was by an intravenous (IV) method.Of note, those clinical trials where efficacy has been demonstrated have been undertaken in the same centre (Mood and Anxieties Disorder Program at the National Institute of Mental Health in Bethesda, MD) with the more recent trials of larger numbers from that centre including individuals that participated in the previous clinical trials. Although beneficial effects have been noted for depressive episodes in both MDD and bipolar disorder, the actual numbers of participants with bipolar disorder has been limited.

Fewer studies have utilised other potential modes of administration for Scopolamine. A previous study of intramuscular scopolamine demonstrated no antidepressant effect whilst one trial of oral scopolamine as an augmentation agent demonstrated an antidepressant effect, albeit this study did not demonstrate a rapid-acting effect as demonstrated in the studies of IV Scopolamine and did not include individuals with bipolar disorder. In addition, oral Scopolamine has very limited bioavailability of ~4 %.Trials relating to administration of Scopolamine utilising a transdermal patch for the management of depressive episodes have yet to be published.

This is a single-site, randomised, double-blind, placebo-controlled, parallel, phase IIb clinical trial. The trial will be sponsored by the National University of Ireland (NUI) Galway and the sponsorship role coordinated by the HRB-Clinical Research facility Galway (CRFG). The site will be University Hospital Galway, Galway and the site activities will also be co-ordinated by the CRFG. Participants will be attending the Galway-Roscommon Mental Health Services, including a specialised bipolar clinic in Galway and referred due to experiencing a depressive episode by their treating clinical team; or patients who have previously attended NUI Galway/HRB-CRFG with an interest to participate/or have participated in research and have indicated a willingness to engage in future research; or patients who approach the research group directly requesting participation.

Trial participants will be adults (both male and female) who have bipolar disorder and are experiencing a depressive episode of at least moderate severity. A diagnosis of bipolar disorder (bipolar 1 or 2 disorder) will be determined by interview with the Structured Clinical Interview for DSM-V (SCID-RV) with severity of the depressive episode assessed using the Hamilton Depression Rating Scale (HDRS) (HDRS ≥14 for study inclusion) at screening.

The primary outcome in this study is the change in severity of depressive symptoms as measured on the Hamilton Depression Rating Scale score (HDRS). Allocating 25 participants to each arm will ensure power ≥85% to detect a 50% lower score on the Hamilton Depression Rating Scale score (HDRS) in the Scopolamine group compared to placebo group. This assumes a loss to follow-up of ≤12%. It is also anticipated that approximately 60 participants will need to be recruited to ensure 50 participants are eligible for randomisation after a placebo run-in.

After a screening Visit (Visit 1); at Visit 2, all participants will receive placebo run-in (100mls of Saline IV). The screening visit (Visit 1) and Visit 2 may occur on the same day. Within 7 days of Visit 2, participants will be randomised (Visit 3) to receive either placebo (n=25) or 4 μg/kg Scopolamine (n=25) IV in 100mls of Saline over 15 minutes at Visits 3 (day 0), 4 (days 2-6) and 5 (days 6-10), with at least 2 days between IV infusions (Visits 2, 3, 4 and 5). Two follow-up visits (Visits 6 and 7) will occur at day 15 (+/-5 days) and day 29 (+/- 7 days).There will be at least 2 days between Visits 5 and 6 and 3 days between Visits 6 and 7. Participants randomised to the placebo group will receive one 15-minute infusion of IV saline,repeated over 3 visits (Visit 3, 4 & 5). The placebo and active comparators will be indistinguishable from each other.

Participants will be randomly assigned to receive either scopolamine or placebo in a 1:1 ratio. Randomly permuted blocks of sizes 4 and 6 will be used to ensure similar numbers of participants in each arm of the trial.

Randomisation will be stratified by the HDRS score at trial entry (a score of <23 indicating a mild-moderate depressive episode and a score ≥23 indicating a severe depressive episode). A validated randomisation system will be used at Visit 3, (after HDRS and Young Mania Rating Scale (YMRS) are completed) to randomise patients to either arm. This centralised system will ensure allocation concealment; preventing blinded trial staff from knowing which treatment group will be allocated. Blocks of randomly varying length will also reduce the predictability of the allocation sequence.

Effectiveness outcomes will be analysed on an intention-to-treat basis for all participants randomised and with available follow-up data as per their randomised allocation. A per-protocol dataset is not well-defined under multiple treatments, here it could reasonably be defined as those participants who either received at least 1, at least 2 or all 3 IV treatments after randomisation. Sensitivity analyses will thus be performed on the primary outcome to assess efficacy of the treatment compared to placebo by incorporating the original allocation of participants and their level of adherence to treatment. This will involve examining the short term-effect of treatment in a longitudinal model and the overall effect of number of IV treatments received at follow-up visits after the final IV treatment.

For the primary effectiveness analysis of the primary outcome, it is expected that pre-randomisation measurements of the HDRS score will be correlated with the scores obtained at Visit 6 of treatment. The mean scores at Visit 6 will be compared across the study arms using an ANCOVA model. The response variable will be the change in HDRS score from Visit 3 to HDRS at Visit 6 including the HDRS score at Visit 3 as a covariate in the model. The addition of stratifying variables and other variables as covariates will be considered as appropriate and specified in the statistical analysis plan. This analysis will increase the power to detect significant differences between the groups. Inverse probability weighting will be applied to the primary outcome analysis. These weights will be derived based on the inverse of the probability of a patient's data being missing given their pre-randomisation measurements. This will ensure the estimate and inference is more representative of all patients randomised, reducing bias in the estimation of the treatment effect due to participants lost to follow-up and missing data.

Inference regarding the treatment effectiveness will focus on the point estimate, confidence interval and p-value for hypothesis confirmation.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each participant must meet all of the following inclusion criteria at Screening (Visit 1) and must continue to fulfil these criteria at Visit 2 to take part in the trial:

1. Diagnosis of Bipolar Disorder according to Diagnostic Statistics Manual (DSM)-V criteria
2. Experiencing an episode of depression of at least moderate severity at Visit 1 (Screening) and Visit 2 based on clinical interview by a trained clinician and a Hamilton Depression Rating Scale (HDRS) score ≥ 14.
3. ≥ 18 years old at Visit 2 (male or female)
4. In the opinion of the Principal Investigator or Sub Investigator's, be able and willing to provide written informed consent and to comply with the requirements of this study protocol.
5. Written informed consent prior to participating in the study
6. Urea and Electrolytes (U&Es), Liver Function Tests (LFTs) and Thyroid Function Tests (TFTs) laboratory tests within acceptable ranges in the previous 4 months of the Screening Visit (Visit 1).

   Placebo run-in inclusion criteria at Randomisation visit (Visit 3):
7. In addition to above, participants must be experiencing an episode of depression of at least mild severity (having previously experienced an episode of moderate depression at Visit 2 with HDRS ≥14), based on clinical interview by a trained clinician and a HDRS score of ≥ 8.

Exclusion Criteria:

Participants who meet any one or more of the following exclusion criteria at Screening (Visit 1) or the Visit 2 will not be eligible to take part in the trial:

1. History of other Axis I diagnosis (including Recurrent Depressive Disorder or Psychotic Disorders such as schizo-affective disorder, conditions that can also present with depressive episodes)
2. History in the three months prior to Visit 2 of alcohol dependence syndrome or substance dependence syndrome.
3. Current use of oral steroid at Visit 1
4. A confirmed diagnosis of dementia
5. A diagnosis of intellectual disability (IQ < 70)
6. Participants with bipolar disorder that are euthymic in the investigators opinion at screening or Visit 2.
7. Participants with bipolar disorder that are hypomanic or manic (Young Mania Rating Scale (YMRS) > 6) at screening or Visit 2.
8. Presence of an established neurological disorder or other serious demyelinating conditions as determined by the treating physician (e.g. space occupying lesion, multiple sclerosis)
9. Current involuntary detention under the Mental Health Act (MHA) 2001 in an acute psychiatric inpatient unit
10. Severity of Bipolar Disorder is such that participation in a clinical trial is not appropriate because of the risk of imminent self-harm (based on clinical note review and review at screening visit by experienced clinician)
11. A history of an allergic reaction or sensitivity to Scopolamine (Hyoscine Hydrobromide). Participants will be asked at the screening visit about any previous treatment with scopolamine (Hyoscine Hydrobromide) to ascertain any previous allergic reaction or sensitivity to this agent.
12. A clinical diagnosis of narrow angle glaucoma, myasthenia gravis, paralytic ileus,pyloric stenosis, toxic megacolon and acute porphyria.
13. Individuals will be excluded from the study if currently prescribed anticholinergic medications, including Physostigmine, Biperiden and Procyclidine. Individuals will additionally be excluded if currently prescribed Tricyclic Antidepressants which are associated with significant anticholinergic properties (e.g. Amitriptyline and Nortriptyline) that are currently causing the participant to experience anticholinergic side effects (e.g. blurred vision, constipation, urinary retention, cognitive difficulties). No individuals will have anticholinergic medications stopped to allow them enter the trial.
14. Bradycardia < 50 bpm, tachycardia > 100bpm or hypotension (systolic BP <90 and / or diastolic BP < 60) prior to IV administration of placebo or Scopolamine
15. A recent history in the last 6 months of symptomatic orthostatic hypotension or syncope.
16. Previous participation in this trial. Participation is defined as randomised. Participation in another trial within 3 months prior to Visit 1. Receipt of any investigational medicinal product (IMP) within 3 months prior to Visit 1.
17. Participants concurrently being administered Electroconvulsive Therapy (ECT).
18. Pregnancy, as determined by a positive urine dipstick at Visits 2, 3, 4, 5, positive blood serum result executed at Visit 2 and confirmed prior to infusion at Visit 3 or participants who are actively breastfeeding (female only).
19. Women of child-bearing potential are defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment. Highly effective contraception methods include:

    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment.
    * Male partner sterilization
    * Combination of any two of the following:

      1. Barrier methods of contraception e.g. Condom
      2. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception
      3. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Women who are considered post-menopausal i.e. amenorrhea at least 12 months or undergone hysterectomy/bilateral oophorectomy
20. Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol

    Placebo run-in exclusion criteria at Randomisation visit (Visit 3):
21. In addition to having completed Visit 2, participants must not be experiencing a hypomanic, or manic episode (YMRS >6).
22. A Serious Adverse Event (SAE) experienced during infusion which required medical intervention and whereby attending physician deemed it inappropriate for the participant to engage in future infusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, County Galway, Ireland

REFERENCES:
- [Background] Belmaker RH. Bipolar disorder. N Engl J Med. 2004 Jul 29;351(5):476-86. doi: 10.1056/NEJMra035354. No abstract available. PMID 15282355
- [Background] Bonner TI, Buckley NJ, Young AC, Brann MR. Identification of a family of muscarinic acetylcholine receptor genes. Science. 1987 Jul 31;237(4814):527-32. doi: 10.1126/science.3037705.
- [Background] Cannon DM, Carson RE, Nugent AC, Eckelman WC, Kiesewetter DO, Williams J, Rollis D, Drevets M, Gandhi S, Solorio G, Drevets WC. Reduced muscarinic type 2 receptor binding in subjects with bipolar disorder. Arch Gen Psychiatry. 2006 Jul;63(7):741-7. doi: 10.1001/archpsyc.63.7.741. PMID 16818863
- [Background] Cannon DM, Klaver JK, Gandhi SK, Solorio G, Peck SA, Erickson K, Akula N, Savitz J, Eckelman WC, Furey ML, Sahakian BJ, McMahon FJ, Drevets WC. Genetic variation in cholinergic muscarinic-2 receptor gene modulates M2 receptor binding in vivo and accounts for reduced binding in bipolar disorder. Mol Psychiatry. 2011 Apr;16(4):407-18. doi: 10.1038/mp.2010.24. Epub 2010 Mar 30. PMID 20351719
- [Background] Davis CE, Applegate WB, Gordon DJ, Curtis RC, McCormick M. An empirical evaluation of the placebo run-in. Control Clin Trials. 1995 Feb;16(1):41-50. doi: 10.1016/0197-2456(94)00027-z. PMID 7743788
- [Background] Davis KL, Berger PA, Hollister LE, Defraites E. Physostigmine in mania. Arch Gen Psychiatry. 1978 Jan;35(1):119-22. doi: 10.1001/archpsyc.1978.01770250121012. PMID 339869
- [Background] Drevets WC, Furey ML. Replication of scopolamine's antidepressant efficacy in major depressive disorder: a randomized, placebo-controlled clinical trial. Biol Psychiatry. 2010 Mar 1;67(5):432-8. doi: 10.1016/j.biopsych.2009.11.021. Epub 2010 Jan 15. PMID 20074703
- [Background] Dwyer JM, Lepack AE, Duman RS. mTOR activation is required for the antidepressant effects of mGluR(2)/(3) blockade. Int J Neuropsychopharmacol. 2012 May;15(4):429-34. doi: 10.1017/S1461145711001702. Epub 2011 Nov 24. PMID 22114864
- [Background] Ellis JS, Zarate CA Jr, Luckenbaugh DA, Furey ML. Antidepressant treatment history as a predictor of response to scopolamine: clinical implications. J Affect Disord. 2014 Jun;162:39-42. doi: 10.1016/j.jad.2014.03.010. Epub 2014 Mar 26. PMID 24767003
- [Background] Ferrari AJ, Stockings E, Khoo JP, Erskine HE, Degenhardt L, Vos T, Whiteford HA. The prevalence and burden of bipolar disorder: findings from the Global Burden of Disease Study 2013. Bipolar Disord. 2016 Aug;18(5):440-50. doi: 10.1111/bdi.12423. PMID 27566286
- [Background] Fournier JC, DeRubeis RJ, Hollon SD, Dimidjian S, Amsterdam JD, Shelton RC, Fawcett J. Antidepressant drug effects and depression severity: a patient-level meta-analysis. JAMA. 2010 Jan 6;303(1):47-53. doi: 10.1001/jama.2009.1943. PMID 20051569
- [Background] Furey ML, Drevets WC. Antidepressant efficacy of the antimuscarinic drug scopolamine: a randomized, placebo-controlled clinical trial. Arch Gen Psychiatry. 2006 Oct;63(10):1121-9. doi: 10.1001/archpsyc.63.10.1121. PMID 17015814
- [Background] Furey ML, Nugent AC, Speer AM, Luckenbaugh DA, Hoffman EM, Frankel E, Drevets WC, Zarate CA Jr. Baseline mood-state measures as predictors of antidepressant response to scopolamine. Psychiatry Res. 2012 Mar 30;196(1):62-7. doi: 10.1016/j.psychres.2012.01.003. Epub 2012 Feb 18. PMID 22349648
- [Background] Furey ML, Drevets WC, Hoffman EM, Frankel E, Speer AM, Zarate CA Jr. Potential of pretreatment neural activity in the visual cortex during emotional processing to predict treatment response to scopolamine in major depressive disorder. JAMA Psychiatry. 2013 Mar;70(3):280-90. doi: 10.1001/2013.jamapsychiatry.60. PMID 23364679
- [Background] GERSHON S, SHAW FH. Psychiatric sequelae of chronic exposure to organophosphorus insecticides. Lancet. 1961 Jun 24;1(7191):1371-4. doi: 10.1016/s0140-6736(61)92004-9. No abstract available. PMID 13704751
- [Background] Gillin JC, Sutton L, Ruiz C, Darko D, Golshan S, Risch SC, Janowsky D. The effects of scopolamine on sleep and mood in depressed patients with a history of alcoholism and a normal comparison group. Biol Psychiatry. 1991 Jul 15;30(2):157-69. doi: 10.1016/0006-3223(91)90170-q. PMID 1655072
- [Background] Janowsky DS, el-Yousef MK, Davis JM, Hubbard B, Sekerke HJ. Cholinergic reversal of manic symptoms. Lancet. 1972 Jun 3;1(7762):1236-7. doi: 10.1016/s0140-6736(72)90956-7. No abstract available. PMID 4113219
- [Background] Janowsky DS. Serendipity strikes again: scopolamine as an antidepressant agent in bipolar depressed patients. Curr Psychiatry Rep. 2011 Dec;13(6):443-5. doi: 10.1007/s11920-011-0239-6. PMID 21976067
- [Background] Kroon JS, Wohlfarth TD, Dieleman J, Sutterland AL, Storosum JG, Denys D, de Haan L, Sturkenboom MC. Incidence rates and risk factors of bipolar disorder in the general population: a population-based cohort study. Bipolar Disord. 2013 May;15(3):306-13. doi: 10.1111/bdi.12058. Epub 2013 Mar 27. PMID 23531096
- [Background] Insel TR, Wang PS. The STAR*D trial: revealing the need for better treatments. Psychiatr Serv. 2009 Nov;60(11):1466-7. doi: 10.1176/ps.2009.60.11.1466. PMID 19880463
- [Background] Khajavi D, Farokhnia M, Modabbernia A, Ashrafi M, Abbasi SH, Tabrizi M, Akhondzadeh S. Oral scopolamine augmentation in moderate to severe major depressive disorder: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2012 Nov;73(11):1428-33. doi: 10.4088/JCP.12m07706. Epub 2012 Oct 16. PMID 23146150
- [Background] Newhouse PA, Sunderland T, Tariot PN, Weingartner H, Thompson K, Mellow AM, Cohen RM, Murphy DL. The effects of acute scopolamine in geriatric depression. Arch Gen Psychiatry. 1988 Oct;45(10):906-12. doi: 10.1001/archpsyc.1988.01800340028004. PMID 3048225
- [Background] Poland RE, Tondo L, Rubin RT, Trelease RB, Lesser IM. Differential effects of scopolamine on nocturnal cortisol secretion, sleep architecture, and REM latency in normal volunteers: relation to sleep and cortisol abnormalities in depression. Biol Psychiatry. 1989 Feb 15;25(4):403-12. doi: 10.1016/0006-3223(89)90193-5. PMID 2930809
- [Background] Popa D, El Yacoubi M, Vaugeois JM, Hamon M, Adrien J. Homeostatic regulation of sleep in a genetic model of depression in the mouse: effects of muscarinic and 5-HT1A receptor activation. Neuropsychopharmacology. 2006 Aug;31(8):1637-46. doi: 10.1038/sj.npp.1300948. Epub 2005 Nov 9. PMID 16292325
- [Background] Porter AC, Bymaster FP, DeLapp NW, Yamada M, Wess J, Hamilton SE, Nathanson NM, Felder CC. M1 muscarinic receptor signaling in mouse hippocampus and cortex. Brain Res. 2002 Jul 19;944(1-2):82-9. doi: 10.1016/s0006-8993(02)02721-x. PMID 12106668
- [Background] ROWNTREE DW, NEVIN S, WILSON A. The effects of diisopropylfluorophosphonate in schizophrenia and manic depressive psychosis. J Neurol Neurosurg Psychiatry. 1950 Feb;13(1):47-62. doi: 10.1136/jnnp.13.1.47. No abstract available. PMID 15405311
- [Background] Yildiz A, Vieta E, Leucht S, Baldessarini RJ. Efficacy of antimanic treatments: meta-analysis of randomized, controlled trials. Neuropsychopharmacology. 2011 Jan;36(2):375-89. doi: 10.1038/npp.2010.192. Epub 2010 Oct 27. PMID 20980991
- [Derived] Miravalles C, Kane R, Rossier AT, Quirke J, Aguilar Macias DA, Alvarez-Iglesias A, Chukwudi K, McDonald C, Cannon DM, Hallahan B. Antidepressant efficacy and safety of scopolamine in individuals with bipolar disorder (SCOPE-BD): A randomized double-blind placebo-controlled trial. J Affect Disord. 2026 Mar 15;397:120888. doi: 10.1016/j.jad.2025.120888. Epub 2025 Dec 16. PMID 41412339
- [Derived] Miravalles C, Kane R, McMahon E, McDonald C, Cannon DM, Hallahan B. Efficacy and safety of scopolamine compared to placebo in individuals with bipolar disorder who are experiencing a depressive episode (SCOPE-BD): study protocol for a randomised double-blind placebo-controlled trial. Trials. 2022 Apr 23;23(1):339. doi: 10.1186/s13063-022-06270-4. PMID 35461262

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 55 participants who consented, 5 were withdrawn pre-randomisation. Three participants were deemed to have HDRS scores below the acceptable eligibility range (<14). A single participant was withdrawn by PI due to being medically (physically) unfit to continue. A single participant withdrew consent due to difficulties with cannulation.
  Fifty participants were randomised into the SCOPE-BD trial.
Groups:
- Scopolamine: Participants randomised to the treatment group will receive one 15-minute IV infusion of Scopolamine (dose 4μg/kg) at 4 visits.
Period: Overall Study
Arm/Group | Placebo | Scopolamine
Started | 24 | 26
Completed | 24 | 23
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Consenting participants who were randomised.
Groups:
- Placebo: The placebo group will receive a 100ml infusion of saline at 4 visits during the study
- Scopolamine: The treatment group will receive a 100ml infusion of Scopolamine (dose 4μg/kg) at 4 visits during the study
- Total: Total of all reporting groups
Arm/Group | Placebo | Scopolamine | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [46 to 57] | 42 [37 to 50] | 48 [39 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 9 | 15 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Hispanic/Latino | 1 | 1 | 2
  White | 23 | 24 | 47
Occupational status [Count of Participants; unit: Participants]
  Employed full-time for pay | 4 | 2 | 6
  Employed part-time for pay | 1 | 5 | 6
  Full-time student | 2 | 1 | 3
  Homemaker | 2 | 1 | 3
  Leave of absence for medical reasons (plan to return to work) | 2 | 4 | 6
  Retired | 3 | 1 | 4
  Unemployed <6 months, but expects to work | 0 | 2 | 2
  Unemployed <6months, does not expect to work | 1 | 1 | 2
  Unemployed >=6months, but expects to work | 2 | 5 | 7
  Unemployed >=6months, does not expect to work | 7 | 4 | 11
Educational status [Count of Participants; unit: Participants]
  College graduate | 11 | 5 | 16
  Graduate professional training (Masters or above) | 6 | 7 | 13
  High school graduate | 3 | 6 | 9
  Junior hhigh school (7th,8th,9th) | 0 | 1 | 1
  Some college or technical school (at least one year) | 3 | 5 | 8
  Some high school (10th,11th) | 1 | 2 | 3
Relationship status [Count of Participants; unit: Participants]
  Divorced | 3 | 3 | 6
  Long-term relationship | 4 | 2 | 6
  Married | 7 | 4 | 11
  Single | 10 | 17 | 27
Socioeconomical status [Count of Participants; unit: Participants]
  Machine operators, semiskilled workers | 3 | 9 | 12
  Major business and professional | 1 | 1 | 2
  Medium business, minor professional, technical | 8 | 6 | 14
  Skilled craftsmen, clerical, sales workers | 7 | 4 | 11
  Unskilled labourers, menial service workers | 5 | 6 | 11
Handedness [Count of Participants; unit: Participants]
  Right-handed | 20 | 23 | 43
  Left-handed | 3 | 1 | 4
  Ambidextrous | 1 | 2 | 3
Psychosis [Count of Participants; unit: Participants] | 10 | 13 | 23
Rapid cycling [Count of Participants; unit: Participants] — Rapid cycling mood disorder is defined as four or more discrete episodes of a mood disorder within 12 months.
  Participants | 2 | 3 | 5
History of involuntary hospitalisation for Bipolar episode [Count of Participants; unit: Participants] | 5 | 10 | 15
History of voluntary hospitalisation for Bipolar episode [Count of Participants; unit: Participants] | 16 | 16 | 32
Smoker [Count of Participants; unit: Participants] | 8 | 9 | 17
Substance use [Count of Participants; unit: Participants] | 9 | 8 | 17
Alcohol use [Count of Participants; unit: Participants] | 7 | 7 | 14
Alcohol dependence [Count of Participants; unit: Participants] | 3 | 5 | 8
Cannabis use [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale Score After Last Treatment
Description: Severity of objective depressive symptoms after the final scheduled treatment (Visit 6) as measured by the Hamilton Depression Rating Scale score. Possible scale range is 0-54, with higher values indicating greater severity of Depression.
Time Frame: Approximately 2 weeks after randomisation (Visit 6)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 24
units on a scale | 12.0 [7.0 to 15.5] | 13.0 [10.8 to 17.0]
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Remission of Depressive Episode After Last Treatment (Visit 6)
Description: Remission of depressive episode after the last IV treatment (measured objectively at Visit 6), defined as occurring when an individual has a Hamilton Depression Rating Scale score <= 7 and a Montgomery and Asberg Depression Scale (MADRS) score <6. The Hamilton Depression Rating Scale possible scale range is 0-54, with higher values indicating greater severity of Depression. The Montgomery-Åsberg Depression Rating Scale Score possible range is 0-60 with higher scores indicating greater severity of Depression.
Time Frame: Approximately 2 weeks after randomisation (Visit 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 24
Participants | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p > 0.9, Fisher Exact

3. Secondary Outcome: Remission of Depressive Episode at Followup (Visit 7)
Description: Remission of depressive episode at followup (measured objectively at Visit 7), defined as occurring when an individual has a Hamilton Depression Rating Scale score <= 7 and a Montgomery and Asberg Depression Scale (MADRS) score <6. he Hamilton Depression Rating Scale possible scale range is 0-54, with higher values indicating greater severity of Depression. The Montgomery-Åsberg Depression Rating Scale Score possible range is 0-60 with higher scores indicating greater severity of Depression.
Time Frame: Approximately 4 weeks after randomisation (visit 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 23
Participants | 4 | 1
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.3, Fisher Exact

4. Secondary Outcome: Response to a Depressive Episode After the Last IV Treatment (Visit 6)
Description: Response to a depressive episode after the last IV treatment (measured at Visit 6) defined as a 50% reduction in Montgomery-Åsberg Depression Rating Scale score at Visit 6 compared to Visit 3. The Montgomery-Åsberg Depression Rating Scale Score possible range is 0-60 with higher scores indicating greater severity of Depression.
Time Frame: Approximately 2 weeks after randomisation (visit 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 24
Participants | 9 | 7
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.5, Chi-squared

5. Secondary Outcome: Remission of Depressive Episode at Followup
Description: Response at Visit 7, defined as a 50% reduction in Montgomery-Åsberg Depression Rating Scale score at Visit 7 compared to Visit 3.
Time Frame: At the time of followup at Visit 7, about 4 weeks after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 23
Participants | 7 | 6

6. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale Score After Last Treatment (Visit 6)
Description: Montgomery-Åsberg Depression Rating Scale Score After Last Treatment (Visit 6). The The Montgomery-Åsberg Depression Rating Scale Score possible range is 0-60 with higher scores indicating greater severity of Depression.
Time Frame: After last treatment (Visit 6), about 2 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 24
units on a scale | 14 [9 to 20] | 16 [10 to 27]
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Total Profile of Mood States Score After Last Treatment (Visit 6)
Description: POMS profile of mood scale is a questionnaire containing 65 words/statements that describe feelings people have. Total Score has range from 0-200 with higher scores indicating greater mood disturbance.
Time Frame: After last treatment (Visit 6), about 2 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 22 | 23
units on a scale | 27 [9 to 51] | 41 [16 to 93]
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Hamilton Depression Rating Scale Score at Followup
Description: Severity of objective depressive symptoms at followup (Visit 7) as measured by the Hamilton Depression Rating Scale score. Possible scale range is 0-54, with higher values indicating greater severity of Depression.
Time Frame: At the time of followup (Visit 7), about 4 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 23
units on a scale | 9 [5 to 14] | 12 [10 to 15]
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale Score at Followup
Description: Montgomery-Åsberg Depression Rating Scale Score at followup (Visit 7). The Montgomery-Åsberg Depression Rating Scale Score possible range is 0-60 with higher scores indicating greater severity of Depression.
Time Frame: At the time of followup (Visit 7), about 4 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 23
units on a scale | 14 [9 to 20] | 16 [10 to 27]

10. Secondary Outcome: Total Profile of Mood States Score at Followup (Visit 7)
Description: as for outcome 7
Time Frame: At the time of followup (Visit 7), about 4 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 22 | 23
units on a scale | 19 [2 to 65] | 61 [30 to 84]
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Introduction of New Antidepressant
Description: Antidepressants medication initiation by a participant due to depressive episodes over the duration of the study (Visit 2 to Visit 7):
  (i) Introduction of a new antidepressant (yes / no)
Time Frame: Between randomisation and time of followup at Visit 7, about 4 weeks duration
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 26
Participants | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p = 0.9, Fisher Exact

12. Secondary Outcome: Increase in Dose of Existing Antidepressant
Time Frame: Between randomisation and time of followup at Visit 7, about 4 weeks duration
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 26
Participants | 4 | 4
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p > 0.9, Fisher Exact

13. Secondary Outcome: Occurrence of Hypo (Manic) Episodes Measured by the Young Mania Rating Scale
Description: Occurrence of hypo (manic) episodes as defined by a score of >6 on the Young Mania Rating Scale during study
Time Frame: Between randomisation and time of followup at Visit 7, about 4 weeks duration
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 26
Participants | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p > 0.9, Fisher Exact

14. Secondary Outcome: Admitted to a Psychiatric Inpatient Unit Due to Depressive Episode
Description: Psychiatric inpatient admission of a participant due to depressive episodes during the trial (Visits 2 to 7)
Time Frame: Between randomisation and time of followup at Visit 7, about 4 weeks duration
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Scopolamine
Number analyzed (Participants) | 24 | 26
Participants | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs Scopolamine; Test type: Superiority; p > 0.9, Fisher Exact

ADVERSE EVENTS:
Time Frame: From randomisation through to study completion, an average of about 4 weeks.
Arm/Group | Placebo | Scopolamine
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 1/24 | 3/26
Other Adverse Events (participants affected / at risk) | 14/24 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Scopolamine (N=26)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Suspected suicide (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Scopolamine (N=26)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 16 (29)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 13 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (5) | 3 (3)
Feeling abnormal (General disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 5 (5)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 8 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Panic reaction (Psychiatric disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 8 (11)
Tension (Psychiatric disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 2 (2)
Thirst (General disorders) | 0 (0) | 3 (5)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT04211961/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT04211961/SAP_001.pdf